CLINICAL TRIAL: NCT06690775
Title: Catalina-2: A Phase 2 Study Evaluating the Efficacy and Safety of TORL-1-23 in Women With Advanced Platinum-Resistant Epithelial Ovarian Cancer (Including Primary Peritoneal and Fallopian Tube Cancers) Expressing Claudin 6
Brief Title: CATALINA-2: A Clinical Study of TORL-1-23 in Platinum-resistant Ovarian Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TORL Biotherapeutics, LLC (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORL123-002; 2024-517190-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal; Fallopian Tube Cancer; Endometrioid Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — pegfilgrastim; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive TORL-1-23 on Day 1 of each 21-day cycle. Additionally, pegfilgrastim will be administered on Day 4 of each 21-day cycle.
  Interventions: Drug: TORL-1-23; Drug: Pegfilgrastim (drug)
- Cohort 2 (Experimental): Participants will receive TORL-1-23 on Day 1 of each 21-day cycle. Additionally, pegfilgrastim will be administered on Day 4 of each 21-day cycle.
  Interventions: Drug: TORL-1-23; Drug: Pegfilgrastim (drug)
- Cohort 3 (Experimental): Participants will receive TORL-1-23 on Day 1 of each 21-day cycle. Additionally, pegfilgrastim will be administered on Day 4 of each 21-day cycle.
  Interventions: Drug: TORL-1-23; Drug: Pegfilgrastim (drug)

INTERVENTIONS:
Drug: TORL-1-23 — 2.4mg/kg intravenous infusion on Day 1 of every 3-week cycle.
  Arms: Cohort 1
Drug: TORL-1-23 — 3.0 mg/kg intravenous infusion on Day 1 of every 3-week cycle.
  Arms: Cohort 2
Drug: TORL-1-23 — 3.4 mg/kg intravenous infusion on Day 1 of every 3-week cycle.
  Arms: Cohort 3
Drug: Pegfilgrastim (drug) — 6.0 mg subcutaneous injection on Day 4 of each cycle.

SUMMARY:
A Phase 2 study to evaluate the safety and efficacy of TORL-1-23 in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. Females ≥18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place) at the time of signing the informed consent.
2. Participants must sign the informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Disease Type:

   * Histologically or cytologically confirmed diagnosis of advanced (unresectable) or metastatic high grade serous ovarian, primary peritoneal (i.e, of primary origin), or fallopian tube cancer. High-grade endometrioid ovarian cancer is permitted for enrollment.
   * Participant's tumor must be positive for CLDN6 expression as defined by the CLDN6 reference laboratory assay. Tumor tissue will be required for submission for CLDN6 testing prior to Cycle 1 Day 1.
   * Participants must have platinum-resistant disease, defined as the following:
   * If participants received only 1 line of platinum-based therapy, they must have completed 4 or more cycles of platinum-containing therapy, must have achieved a CR or PR, and progressed >3 months but ≤6 months after the last dose of platinum.
   * Participants who have received more than 1 line of platinum- based therapy must have progressed on or within 6 months after the last dose of platinum.
   * NOTE: This should be calculated from the date of the last administered dose of platinum therapy to the date of the radiographic imaging showing progression (per RECIST v1.1).
   * Participants who are platinum-refractory during front-line treatment are excluded.
   * Participants must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy, and for whom single- agent therapy is appropriate as the next line of treatment. Study rules for evaluation of number of prior systemic lines of therapy:
   * Adjuvant ± neoadjuvant is considered one line of therapy
   * Maintenance therapy (eg, bevacizumab or PARP inhibitors) will be considered part of the preceding line of therapy (ie, not counted independently)
   * Therapy changed due to toxicity in the absence of progression will be considered part of the same line (ie, not counted independently)
   * Hormonal therapy will not be counted as a separate line of therapy
4. Measurable disease, per RECIST v1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
6. Adequate organ function, based on the following laboratory values:

   * ANC: ≥1,500/mcL
   * Platelets: ≥100,000/mcL without transfusion within 4 weeks of first dose
   * Hemoglobin: 9 g/dL with transfusion or EPO support up to 14 days before eligibility assessment
   * Measured or calculated creatinine clearance with a validated formula*: ≥30 mL/min
   * Serum total bilirubin: ≤1.5 X ULN (participants with known Gilbert disease or liver metastases who have serum bilirubin level ≤3×ULN may be enrolled
   * AST (SGOT) and ALT (SGPT): ≤3 X ULN (participants with active liver metastases who have ALT/AST ≤5 X ULN may be enrolled)
   * Albumin: ≥2.5 g/dL
   * ECG: 12-Lead ECG with normal tracing or non-clinically significant changes that do not require medical intervention and QTcF interval

     * 470 msec and without history of Torsades des Pointes or other symptomatic QTc abnormality.
7. Participants of childbearing potential must have a negative serum pregnancy test within 72 hours before starting study drug treatment. The serum pregnancy test must be negative for the participant to be eligible.
8. Participants must agree to use a highly effective birth control method from the time of the first study drug treatment through 7 months after the last study drug treatment, or be of nonchildbearing potential.
9. Participants must agree not to donate eggs from the first study drug treatment through 7 months after the last study drug treatment.
10. Participants must agree to not breastfeed from the first dose of study treatment through 90 days after the last dose of study treatment.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has not recovered [recovery is defined as National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, Grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
2. Participants with clear cell, mucinous, sarcomatous (including carcinosarcoma), mixed histology, or low-grade, borderline ovarian tumors or non-epithelial ovarian cancers.
3. Participants with primary platinum-refractory ovarian, primary peritoneal (i.e. of primary origin) or fallopian tube cancer, defined as disease that did not respond to or has progressed within 3 months of the last dose of first line platinum-containing chemotherapy.
4. Received prior chemotherapeutic, investigational, radiotherapy, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of TORL-1-23. There is no waiting period required for stereotactic radiosurgery.
5. Prior treatment with a CLDN6-targeting agent or an MMAE-containing ADC.
6. Progressive or symptomatic brain metastases. Brain metastases that have been radiated, are asymptomatic, and on a stable or decreasing dose of steroids are allowed. Leptomeningeal disease is excluded.
7. Grade 2 or greater peripheral neuropathy.
8. History of non-infectious pneumonitis/ILD within 6 months of first dose of study drug.
9. Participants must not be considered a high medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
10. History of significant cardiac disease:

    1. Congestive heart failure >New York Heart Association class 2 within last year
    2. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
    3. Myocardial infarction less than 6 months before start of study drug
    4. Anti-arrhythmic therapy (beta blockers are permitted)
    5. Any unstable ischemic disease or untreated arrhythmia
11. Known history of myelodysplastic syndrome or acute myeloid leukemia.
12. History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. Participants with malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ of the breast are not excluded.
13. Uncontrolled infection; active, clinically serious infections (CTCAE Grade >2).
14. Participants with seizure disorder requiring medication.
15. Known hypersensitivity or intolerance to any of the study drugs, study drug classes, or excipients in the formulation.
16. History of having an allogeneic bone marrow or organ transplant.
17. Any condition (concurrent disease, infection, or comorbidity) that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator.
18. Participants who are taking any drugs that are strong inducers and/or strong inhibitors of CYP3A4 enzymes.
19. Participants who are taking any drugs that are inhibitors of P-glycoprotein.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 230 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of TORL-1-23 as a monotherapy in women with advanced PROC expressing CLDN6 | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 40 months
  Objective Response Rate (ORR) per RECIST v1.1 by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
Duration of Response (DOR) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 40 months
  To assess additional efficacy outcome measures of TORL-1-23 per RECIST v1.1 by Blinded Independent Central Review (BICR) and investigator assessment
Objective Response Rate (ORR) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 40 months
  To assess additional efficacy outcome measures of TORL-1-23 per RECIST v1.1 by investigator assessment
Progression-free Survival (PFS) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 40 months
  To assess additional efficacy outcome measures of TORL-1-23 per RECIST v1.1 by Blinded Independent Central Review (BICR) and by investigator assessment
Overall Survival (OS) | From time of consent until death or completion of study (Study duration is approximately 40 months)
  To assess additional efficacy outcome measures of TORL-1-23
Incidence and severity of AEs and clinical laboratory abnormalities per CTCAE v5.0 | From informed consent until 30 days after the last dose of study treatment, approximately 24 months (each cycle is 21 days)
  To assess the safety and tolerability of TORL-1-23
CA-125 response per Gynecological Cancer Intergroup (GCIG) criteria | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 40 months
  To assess the pharmacodynamic effects of TORL-1-23

CONTACTS AND LOCATIONS:
Locations (66):
- United States (26):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - SCRI - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Providence St. Jude Medical Center, Fullerton, California
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - SCRI - Sansum Clinic, Santa Barbara, California
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - SCRI - Maryland Oncology Hematology, P.A., Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - SCRI - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Duke Cancer Center, Durham, North Carolina
  - The James Cancer Hospital and Solove Research Institute - Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center at the University of Oklahoma, Oklahoma City, Oklahoma
  - SCRI - Northwest Cancer Specialists, P.C., Portland, Oregon
  - SCRI - Alliance Cancer Specialists, PC, Doylestown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI - Texas Oncology, Fort Worth, Texas
  - SCRI - Virginia Oncology Associates, Norfolk, Virginia
- Australia (5):
  - Monash Medical Centre, Clayton, Melbourne
  - Blacktown Hospital, Blacktown, New South Wales
  - Icon Cancer Centre Chermside, Chermside, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Linear Clinical Research, Perth, Western Australia
- Austria (3):
  - Medizinische Universitat Landeskrankenhaus Graz, Graz, Styria
  - Universitatsklinik Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz, Linz, Upper Austria
- Belgium (4):
  - Antwerp University Hospital (UZA), Edegem, Antwerp
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Leuven, Leuven, Flemish Brabant
  - CHU Liège, Liège, Wallonia
- Canada (8):
  - BC Cancer - Abbotsford, Abbotsford, British Columbia
  - British Columbia Cancer Agency (BC Cancer, part of the Provincial Health Services Authority), Vancouver, British Columbia
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre - University Health Network (UHN), Toronto, Ontario
  - Hospital Maisonneuve Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre (MUHC) - Royal Victoria Hospital, Montreal, Quebec
- France (3):
  - Centre Leon Berard, Lyon, Auvergne- Rhôn-Alpes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Pays de la Loire Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (3):
  - Universitatsklinikum Heidelberg, Heidelberg, Baden-Wurttenberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
- Ireland (2):
  - Start Dublin - Mater Misericordiae University Hospital, Dublin, Leinster
  - St. James Hospital, Dublin, Leinster
- Italy (4):
  - IRCCS Giovani Paolo II - Instituto Oncologico, Bari, Apulia
  - Humanitas San Pio X, Milan, Milano
  - Nuovo Ospedale di Prato S Stefano, Prato, Prato
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Rome
- Singapore (3):
  - National University Cancer Institute, Singapore, Singapore
  - National Cancer Centre, Singapore, Singapore
  - Curie Oncology (Farrer), Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul, Gwanak-gu
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seocho-Gu
  - Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-Gu
  - Asan Medical Center, Seoul, Songpa-Gu
- Institut Catalá d'Oncologia de Girona, Girona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided